CLINICAL TRIAL: NCT05505994
Title: A Multi-center, Randomized, Double-Blind, Active-controlled, Phase 3, Therapeutic Confirmatory Study and Open-Label Extension Study to Evaluate the Efficacy and Safety of DWP16001 Add-on to Metformin in Patients With Type 2 Diabetes Mellitus Inadequately Controlled on Metformin
Brief Title: The Efficacy and Safety of DWP16001 in Combination With Metformin in T2DM Patients Inadequately Controlled on Metformin
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP16001304_CN
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Disease; Endocrine System Diseases
Keywords: Dapagliflozin; Sodium-Glucose Transporter 2 Inhibitors; Molecular Mechanisms of Pharmacological Action; Hypoglycemic Agents; Physiological Effects of Drugs
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Glucose Metabolism Disorders; Metabolic Diseases; Endocrine System Diseases | interventions — Enavogliflozin; dapagliflozin

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 1: Double-blind Part 2: Open label
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): DWP16001 A mg, Dapagliflozin placebo
  Interventions: Drug: DWP16001; Drug: Dapagliflozin Placebo
- Control group (Active Comparator): DWP16001 A mg placebo, Dapagliflozin
  Interventions: Drug: Dapagliflozin; Drug: DWP16001 Placebo

INTERVENTIONS:
Drug: DWP16001 — DWP16001 A mg tablet
  Other Names: DWP16001 tablet
  Arms: Study group
Drug: Dapagliflozin — Dapagliflozin tablet
  Other Names: Dapagliflozin tablet
  Arms: Control group
Drug: DWP16001 Placebo — DWP16001 Placebo tablet
  Other Names: DWP16001 Placebo tablet
  Arms: Control group
Drug: Dapagliflozin Placebo — Dapagliflozin Placebo tablet
  Other Names: Dapagliflozin Placebo tablet
  Arms: Study group

SUMMARY:
Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of DWP16001 in Combination with Metformin in Patients With Type 2 Diabetes Mellitus who Have Inadequate Glycemic Control on Metformin Alone.

DETAILED DESCRIPTION:
A Multi-center, Randomized, Double-Blind, Active-controlled, Phase 3, Therapeutic Confirmatory Study to Evaluate the Efficacy and Safety of DWP16001 in Combination with Metformin in Patients With Type 2 Diabetes Mellitus who Have Inadequate Glycemic Control on Metformin Alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with T2DM aged 18 to 80 years
2. Subjects who have received metformin alone at a fixed dose for the last 8 weeks and has 7% ≤ HbA1c ≤ 10.5%
3. Subjects with BMI of 20-45 kg/m2
4. Subjects who voluntarily decided to participate and provided written consent after being told of the objectives, method, and effects of this study

Exclusion Criteria:

1. Subjects with current or history of hypersensitivity to the IP of this study, metformin or drugs of the same class and their components (e.g., history of hypersensitivity to biguanide or SGLT2 inhibitors)
2. Diabetic ketoacidosis, diabetic coma or precoma within the past year
3. Urinary tract infections or genital infections within
4. Uncontrolled hypertension (SBP > 180 mmHg or DBP > 110 mmHg)
5. eGFR < 60 mL/min/1.73 m2
6. Severe heart failure (NYHA class III/IV)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 340 (Actual)
Dates: Start 2022-09-28 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in HbA1c | at 24 weeks
  Change in HbA1c (%) is assessed with the values measured at the central laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Linong Ji, Dr., Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided